CLINICAL TRIAL: NCT01298752
Title: The Efficacy and Safety of Mapracorat Ophthalmic Suspension, 3% in Subjects for the Treatment of Ocular Inflammation Following Cataract Surgery
Brief Title: Mapracorat Ophthalmic Suspension, 3% for the Treatment of Ocular Inflammation Following Cataract Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated.
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 664
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Inflammation; Pain; Cataract
MeSH Terms: conditions — Inflammation; Pain; Cataract | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mapracorat (Experimental): Mapracorat ophthalmic suspension
  Interventions: Drug: Mapracorat
- Vehicle (Placebo Comparator): Vehicle of mapracorat ophthalmic suspension
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Mapracorat — Mapracorat ophthalmic suspension 3%, one drop in post-operative study eye once daily (QD) for 2 weeks.
  Other Names: BOL-303242-X
  Arms: Mapracorat
Drug: Vehicle — Vehicle of mapracorat ophthalmic suspension, one drop in post-operative study eye once daily (QD) for 2 weeks.
  Arms: Vehicle

SUMMARY:
The objective of this study is to compare the safety and efficacy of Mapracorat Ophthalmic Suspension, 3% to vehicle for the treatment of postoperative inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are candidates for routine, uncomplicated cataract surgery.
* Subjects must be willing to wait to undergo cataract surgery on the fellow eye until after the study has been completed.

Exclusion Criteria:

* Subjects who are expected to require treatment with any systemic or ocular (either eye) drugs specified in the protocol during the 18 days following cataract surgery or any systemic or ocular corticosteroids within 14 days prior to cataract surgery.
* Subjects who have known hypersensitivity or contraindication to the study drug(s) or their components.
* Subjects who have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mapracorat | Vehicle
Started | 120 | 57
Completed | 77 | 31
Not Completed | 43 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mapracorat | Vehicle | Total
Number analyzed (Participants) | 120 | 57 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.72) | 63.2 (12.29) | 65.4 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 30 | 105
  Male | 45 | 27 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells.
Description: Anterior chamber (AC) cells were assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
Time Frame: 8 days
Population: Randomized participants were included without imputation of missing data at 8 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 114 | 54
Participants | 9 | 6

2. Primary Outcome: Percentage of Participants With Grade 0 Pain
Description: Ocular pain was defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. The scores ranged from 0=None to 5=Severe, where higher scores indicated worse pain.
Time Frame: 8 days
Population: Randomized participants were included without imputation of missing data at 8 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 114 | 54
Participants | 65 | 27

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | Mapracorat | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/57
Other Adverse Events (participants affected / at risk) | 5/120 | 6/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mapracorat (N=120) | Vehicle (N=57)
Eye pain (Eye disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.